CLINICAL TRIAL: NCT06271148
Title: Career and Lifestyle Among Female Surgeons in Jordan
Status: Completed | Type: Observational
Sponsor: Mohammad Abu-Jeyyab (Other)
Responsible Party: Sponsor-Investigator, Mohammad Abu-Jeyyab, General Surgery Department, Mutah university, Mutah University
Organization: Mutah University (Other)
Other Study IDs: Mutah University; Myah REC/133/2023 (Registry Identifier: Mutah university school of medicine)
Record Dates: First submitted 2024-02-02; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Surgery; Lifestyle
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female surgeons: Female surgeons
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — We made multiple interviews with randomly selected surgical candidates

SUMMARY:
A study conducted to evaluate the female surgeons in Jordan from different lifestyle

DETAILED DESCRIPTION:
A study conducted to evaluate the female surgeons in Jordan from different lifestyle challenges

ELIGIBILITY:
Inclusion Criteria:

* female General surgery practitioners Lives in Jordan

Exclusion Criteria:

* males Other surgical specialists Outside Jordan

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females
Study Population: Female in General Surgery practice
Sampling Method: Probability Sample
Enrollment: 224 (Actual)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-12-17 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Career and Lifestyle Among Female Surgeons in Jordan | 5 years
  Career Challenges and Lifestyle Among Female Surgeons in Jordan
Working Hours | 5 years
  Working hours
Sex Bias | 5 years
  sex bias
inadequate mentorship | 5 years
  inadequate mentorship
having 30 days of leave | 5 years
  having 30 days of leave
salary | 5 Years
  salary

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Abu-Jeyyab, Principal Investigator — Mutah University
Locations (1):
- Mutah University, Qīr Moāv, Jordan

IPD SHARING:
Plan to Share IPD: Undecided